CLINICAL TRIAL: NCT01684813
Title: A Randomized Study With Loading Dose of Prasugrel Opposed to the Standard Dose of Clopidogrel in Type 2 Diabetic Patients in Acute Coronary Syndrome, Revascularized Through Drug-eluting Stent.
Brief Title: VERifynow in DIabetes Non-responsiveness: a Study on Switching From Clopidogrel to Prasugrel
Acronym: VERDI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VERDI study
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes Mellitus Type II; Acute Coronary Syndrome
Keywords: Diabetes mellitus.; Acute coronary syndrome.; Percutaneous coronary intervention.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Acute Coronary Syndrome; Diabetes Mellitus | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel (Active Comparator): This group will receive after PCI the standard dose of clopidogrel, a daily dose of 75 mg.
  Interventions: Drug: Clopidogrel
- Prasugrel (Experimental): This group will receive after PCI a loading dose of 60 mg prasugrel (6 x 10 mg tablets) followed by a daily dose of prasugrel (10 mg tablet).
  Interventions: Drug: Prasugrel.

INTERVENTIONS:
Drug: Prasugrel. — Patients in this group will receive a loading dose of 60 mg prasugrel (6 x 10 mg tablets) followed by at least dose of 10 mg prasugrel (1 x 10 mg tablet). Beyond the second day after PCI, these patients will receive double antiaggregation therapy according to their physician´s criteria.
  Other Names: Efient, Eli Lilly
  Arms: Prasugrel
Drug: Clopidogrel — Patients in this group will receive the standard dose of clopidogrel, a daily dose of 75 mg. Beyond the second day post-PCI, these patients will receive double anti aggregation therapy according to their physician's criteria.
  Other Names: Agrelan
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to determine if, in type 2 diabetic patients undergoing treatment with PCI and a stent, who fail to respond to normal doses of clopidogrel, a loading dose of 60 mg of prasugrel followed by 10 mg once daily is superior to the standard dose of 75 mg of clopidogrel in achieving greater than 50% inhibition of platelet aggregation at 24-36 hours of treatment.

DETAILED DESCRIPTION:
The VERDI study consists on a randomized, mono-center study comparing the treatment plan of a loading dose of prasugrel as opposed to the standard dose in type 2 diabetic patients, who suffer acute coronary syndrome, revascularized through an invasive percutaneous strategy with a stent. The aim of this study is to determine if, in type 2 diabetic patients undergoing treatment with PCI and a stent, who fail to respond to normal doses of clopidogrel, a loading dose of 60 mg of prasugrel followed by 10 mg once daily is superior to the standard dose of 75 mg of clopidogrel in achieving greater than 50% inhibition of platelet aggregation at 24-36 hours of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic patients with acute coronary syndrome with non-ST segment elevation who are undergoing a percutaneous coronary intervention (PCI) with a coronary stent.
2. Patients who are non-responsive on the platelet anti-aggregation test with standard doses of clopidogrel will be randomized.
3. Participants must sign an informed consent document.

Exclusion Criteria:

1. Age <18 years or >80 years.
2. Patients with acute coronary syndrome with ST segment elevation.
3. Pregnancy previous to or during the study.
4. The use of oral anticoagulants in the last 10 days with an INR >1.5 or who plan to use them during the follow-up period (1 year).
5. Antithrombotic treatment with GP IIb/IIIa inhibitors.
6. Contraindication for the use of prasugrel and/or clopidogrel and/or aspirin:

   * Antecedents of pharmacologic allergy to thienopyridine derivatives or aspirin.
   * Antecedents of clinically significant or persistent thrombocytopenia or neutropenia.
7. Active bleeding or significant increase of risk of hemorrhage such as severe hepatic insufficiency, peptic ulcer present, proliferative diabetic retinopathy, antecedents of severe systemic bleeding, gastrointestinal bleeding, macrohematuria, intraocular hemorrhage, hemorrhagic stroke, or intracranial bleeding), or other antecedents of bleeding diathesis or coagulopathy.
8. Patients with previous TIA or CVA.
9. Patients weighing <60 Kg.
10. Hemoglobin <10.5 g/dl, or Hematocrit <30%.
11. Severe left ventricular systolic dysfunction, EF <35%.
12. Renal insufficiency with creatinine levels >2 mg/dl.
13. Previous inclusion of the patient in another study.
14. Treatment in research (medication or device) in the last 30 days prior.
15. Medical, geographical, or social factors that would make participation in the study impractical, such as the incapacity to provide written informed consent and to understand the complete meaning of informed consent, or the refusal of the patient to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of patients who achieve inhibition of platelet aggregation greater that 50% | 24 to 36 hours post-PCI
  The principal objective is to determine whether in type 2 diabetic patients who are non-responsive to clopidogrel at habitual doses and who receive treatment through percutaneous coronary intervention (PCI) with a stent, a treatment plan with a loading dose of prasugrel (60 mg) followed by 1 cp (10 mg) once a day, is superior to a standard dose of 75 mg clopidogrel in achieving greater than 50% inhibition of platelet aggregation at 24-36 hours of treatment.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 30 days
  To evaluate the safety of treatment with prasugrel in comparison with the standard treatment with clopidogrel in terms of the appearance of secondary effects (severe bleeding, thrombocytopenia, neutropenia, gastrointestinal changes, thrombotic thrombocytopenic purpura).
Number of patients who die or present the combined endpoint of cardiovascular death, MI or recurrent ischemia as a measure of efficacy. | 30 days.
  To assess the results in different sub-groups and analyze the combined endpoint of cardiovascular death, MI or recurrent ischemia at 30 days.
Number of participants who are non-responsiveness to antiaggregation therapy as a measure of efficacy | 30 days.
  To analyze the characteristics of patients who are non-responsive to anti-aggregation therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Seville, Spain

REFERENCES:
- [Derived] Cubero Gomez JM, Acosta Martinez J, Mendias Benitez C, Diaz De La Llera LS, Fernandez-Quero M, Guisado Rasco A, Villa Gil-Ortega M, Sanchez Gonzalez A. VERifyNow in DIabetes high-on-treatment platelet reactivity: a pharmacodynamic study on switching from clopidogrel to prasugrel. Acta Cardiol. 2015 Dec;70(6):728-34. doi: 10.2143/AC.70.6.3120187. PMID 26717223